CLINICAL TRIAL: NCT05743972
Title: Contrast-Enhanced Ultrasound vs Conventional US-guided Percutaneous Needle Biopsy for Pancreatic Diseases: Prospective Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: xiao-yan xie (Other)
Responsible Party: Sponsor-Investigator, xiao-yan xie, M.D., First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BZhuang
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEUS-guided core biopsy group (Experimental)
  Interventions: Diagnostic Test: Contrast-enhanced ultrasound-guided core biopsy
- US-guided core biopsy group (Active Comparator)
  Interventions: Diagnostic Test: Conventional ultrasound-guided core biopsy

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced ultrasound-guided core biopsy — Core biopsy was used to collect samples for pancreatic diseases under contrast-enhanced ultrasound-guided.
  Arms: CEUS-guided core biopsy group
Diagnostic Test: Conventional ultrasound-guided core biopsy — Core biopsy was used to collect samples for pancreatic diseases under conventional ultrasound-guided.
  Arms: US-guided core biopsy group

SUMMARY:
According to previous studies, contrast-enhanced ultrasound (CEUS) -guided Core Biopsy(GB) could improve the diagnosis of biopsy in liver and other superficial mass compared to conventional US-GB. The purpose of this randomized trial is to estimate whether CEUS-GB achieve excellent diagnostic value to conventional US-GB in percutaneous biopsy for pancreatic diseases.

DETAILED DESCRIPTION:
The patients with pancreatic diseases who need receive percutaneous biopsy were randomized with 1:1 ratio into undergo CEUS-GB group and conventional US-GB group.The aims include:

Comparison the diagnostic accuracy rate between CEUS and US group. Comparison the diagnostic specificity, sensitivity and complication rate between CEUS and US group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, WHO/ECOG scores <2;
* Radiographic examination reveal focal pancreatic lesions;
* No history of local treatment for pancreatic lesions, systemic chemotherapy, targeting, immunotherapy, etc;
* Normal organ function, including the following criteria:

  1. Routine blood test: Hb≥80 g/L; PLT≥50×109/L;
  2. Coagulation function test: PT<20s.

Exclusion Criteria:

* The lesions could not be shown by ultrasound and contrast-enhanced ultrasound;
* Allergic to ultrasound contrast agent;
* Cardiovascular and cerebrovascular diseases, liver, kidney and lung failure with significant clinical symptoms;
* History of unexplained bleeding, severe anemia, bleeding tendency or uncorrected coagulopathy;
* Combined with active infection;
* Massive ascites;
* Patients or family members do not agree to enter the study;
* Pregnant or lactating women;
* The investigator considers that there are any other factors that may be inappropriate for inclusion or affect the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy rate | 6 month
  Diagnostic accuracy rate was defined as the proportion of patients who reached successful diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No